CLINICAL TRIAL: NCT04212195
Title: Cohort Research On Wilson's Disease: Genetic Determinants and Biomarker Discovery for Neurological Involvement
Brief Title: Cohort Research on Wilson's Disease
Acronym: CROWD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 18/0200
Record Dates: First submitted 2019-12-18; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Wilson's Disease
Keywords: Genetic modifiers; Biomarkers
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — High-Throughput Nucleotide Sequencing; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva (part 1). Urine, blood and, in a subset, cerebrospinal fluid (part 2).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part 1: Genetic determinants (n=500)
  Interventions: Genetic: Next generation sequencing
- Part 2: Biomarker discovery (n=40)
  Interventions: Diagnostic Test: Imaging and fluid biomarkers

INTERVENTIONS:
Genetic: Next generation sequencing — Saliva samples
  Groups: Part 1
Diagnostic Test: Imaging and fluid biomarkers — Magnetic resonance imaging of the brain and urine, blood and cerebrospinal fluid sampling
  Groups: Part 2

SUMMARY:
Wilson's disease (WD) is an inherited disorder that causes abnormal copper accumulation in the brain and/or liver. Some people develop neurological or psychiatric symptoms whereas other develop liver disease. The reasons for this are unclear but genetic factors are likely to contribute. Current treatment, using copper-binding medications, is required lifelong. Some respond well but others suffer debilitating side-effects or deteriorate despite treatment, leading to disability or the need for liver transplantation.

In the first part of this study the main aim is to identify genetic factors that determine whether someone with a diagnosis of WD will develop neurological involvement or not. The investigators will invite 500 adults with WD across the UK to take part. Participants will be asked to complete an online questionnaire and provide a saliva sample for genetic testing using a collection kit sent via post. Identifying these genetic factors would significantly advance our understanding of the disease and may provide new targets for drug discovery or help guide more personalised approaches to treatment.

In the second part of this study the main aim is to develop new ways to monitor the effect of WD on the brain using tests. Copper levels in blood and urine, currently used to monitor the disease, are unreliable and do not necessarily reflect ongoing brain damage. The role of MRI scans, cerebrospinal fluid tests or other measures of brain damage, commonly used in other neurological disorders, is unclear. The investigators will therefore follow a group of 40 patients using clinical assessments and a combination of neurological tests, including novel imaging and laboratory techniques, over 24 months. Developing new approaches to monitoring the effect of WD on the brain will enable better prevention of neurological disability and be essential for demonstrating the effectiveness of new treatments, such as gene therapy, in clinical trials in the future.

ELIGIBILITY:
Inclusion Criteria (part 1 and part 2):

* Diagnosed with Wilson's disease
* Age 16 years or over
* Living in the UK

Exclusion Criteria (part 2):

* Participant has another medical or psychiatric illness that would interfere in completing assessments
* Participant is pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Secondary care
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2021-12-06 (Estimated); Study Completion 2021-12-06 (Estimated)

PRIMARY OUTCOMES:
Clinical phenotype | Questionnaire responses will be collected over two years.
  Responses to online questionnaires for the first part of the study will be used to the determine the presence or absence of neurological symptoms.
Unified Wilson's Disease Rating Scale (UWDRS) | This assessment will be performed at two research visits 12-18 months apart.
  Participants in the second part of the study will be assessed at research visits using this scale (0-320)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Warner, Principal Investigator — UCL Queen Square Institute of Neurology
Locations (11):
- United Kingdom (11):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff and Vale University Health Board, Cardiff
  - King's College Hospital NHS Foundation Trust, London
  - National Hospital for Neurology and Neurosurgery, London
  - Royal Free London NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Salford Royal NHS Foundation Trust, Salford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield